CLINICAL TRIAL: NCT01615107
Title: Comparison Between the Use of Standard Oxytocin Induction Protocol and the Double-balloon Catheter Device With Concurrent Oxytocin
Brief Title: Premature Rupture of Mambrane and Unfavourable Cervix
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0013-12-HYMC
Record Dates: First submitted 2012-04-23; First posted 2012-06-08 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-04

CONDITIONS: Cervix; Insufficient Dilatation in Labor
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GROUP 1: Oxytocin infusion alone (Experimental): GROUP 1: Oxytocin infusion alone
  Interventions: Drug: PITOCIN
- double balloonand oxytocin (Experimental): insertion of the double balloon and oxytocin
  Interventions: Device: COOK RIPENENIG BALLOON+PITOCN; Other: double balloonand oxytocin; Other: ballon and oxytocin; Procedure: double balloonand and oxytocin

INTERVENTIONS:
Device: COOK RIPENENIG BALLOON+PITOCN — GROUP 2: insertion of the double balloon device and concurrent oxytocin administration.
  Other Names: BALLOON+PITOCN
  Arms: double balloonand oxytocin
Drug: PITOCIN — : Oxytocin infusion alone (Standard Protocol
  Other Names: Oxytocin infusion alone
  Arms: GROUP 1: Oxytocin infusion alone
Other: double balloonand oxytocin — balloonand oxytocin
  Other Names: balloonand oxytocin
  Arms: double balloonand oxytocin
Other: ballon and oxytocin — double- balloon catheter device with concurrent oxytocin
  Other Names: balloon catheter device with concurrent oxytocin
  Arms: double balloonand oxytocin
Procedure: double balloonand and oxytocin — balloon catheter device with concurrent oxytocin
  Other Names: balloon catheter device with concurrent oxytocin
  Arms: double balloonand oxytocin

SUMMARY:
The paucity of published data concerning the issue of mechanical labor induction in the setting of Term PROM has led us to undertake the present clinical trial. This study is designed to compare the efficacy and safety of the standard Oxytocin induction protocol with the double-balloon catheter device with concurrent oxytocin administration in patients with Term PROM and unfavorable cervical conditions.

DETAILED DESCRIPTION:
This will be a prospective randomised trial. Two hundred pregnant women with term PROM and an unfavourable cervix (Bishop Score ≤ 4) are expected to be entered into the study (see statistical analysis below).

All eligible women will be presented with the study protocol by a study coordinator. Women interested in participating will read and sign the informed consent. Subsequently, the following screening medical procedures will be completed: medical and gynecological history, physical and vaginal examination, ultrasonography to: (i) Confirm fetal vertex presentation, (ii) Exclude placenta previa and (iii) Assess cervical length and posterior cervical angle. (iv) Asses bio-physical profile score

A non-stress test will be performed in order to monitor:

1. The fetal heart pattern for the presence or absence of decelerations and
2. The presence of uterine contractions. All women will undergo a pelvic examination by a staff member to obtain an initial Bishop score.

If the patient will be determined eligible for study entry, and following the informed consent, randomisation into the following groups will take place:

GROUP 1: Oxytocin infusion alone (Standard Protocol). GROUP 2: insertion of the double balloon device and concurrent oxytocin administration.

GROUP 3: Expectant management

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed to be pregnant with PROM at > 34 week
2. Found to have a Bishop score of 4 points or less.
3. Diagnosed as having a singleto
4. Willingness to comply with the protocol for the duration of the study.
5. Have signed an informed consent.

Exclusion Criteria:

1. Any contraindication for a vaginal deliver
2. Regular uterine contractn
3. Evidence of chorio-amonitis
4. Previous cesarean section or presence of any uterine scar.
5. Suspected placental abruption or presence of a significant hemorrhage.
6. Non-reassuring fetal statu

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
PPROM/PROM to delivery interval | 3year
  Time from rupture of mambrane to delivery
  From hospitalization until delivery

CONTACTS AND LOCATIONS:
Overall Officials: Elad Mei-Dan, DR, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264